CLINICAL TRIAL: NCT03677700
Title: Evaluation of Inflammation of the Anterior Segment by Laser Flashmeter in Patients Having Undergone Surgery of the Posterior Segment (Vitrectomy or Preindentation) During the First Postoperative Year. (FLAVIC)
Acronym: FLAVIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3043_FLAVIC
Record Dates: First submitted 2018-05-17; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-05

CONDITIONS: Inflammation Eye
Keywords: vitrectomy; cryoindentation
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Laser Flare Meter — Measurement of the inflammation of the operated eye and the fellow eye before the surgery and at each post-surgery visit: D7, M1, M2, M3, M6, M12

SUMMARY:
Observational study, monocentric, prospective, descriptive and comparative (eye operated vs fellow eye).

DETAILED DESCRIPTION:
After surgery by vitrectomy or preindentation, an anti-inflammatory treatment is conventionally prescribed for a duration of 1 month. However, frequently, during the post-operative control at one month, there may be signs of ocular inflammation or symptoms of discomfort justifying the prolongation of post-operative treatment. A 2012 study evaluated post-operative flare follow-up in 22 vitrectomized patients for retinal detachment, and showed a significantly higher flare 3 months after surgery, compared to the other eye and pre-surgery value.

In this study, the investigators wish to study postoperative inflammation in patients operated for posterior segment ocular surgery (vitrectomy or preindentation) measured by laser flashmeter on a follow-up of one year.

ELIGIBILITY:
Inclusion Criteria:

* Major patient,
* Operation of vitrectomy or preindentation in the ophthalmology department of Rennes University Hospital for one of the following reasons:
* Retinal detachment, rhegmatogenous or not
* Combined surgery
* Membrane peeling
* Macular hole
* Optically targeted vitrectomy (Terson's syndrome, intravitreous haemorrhage)
* Covered by a health insurance system,
* Having received information on the protocol and not having expressed opposition to participating in the study

Exclusion Criteria:

* Vitrectomy for endophthalmitis or posterior uveitis,
* Patient with vitreoretinal proliferation (grade B and C),
* Pregnant or nursing woman,
* Major patient subject to legal protection (safeguard of justice, guardianship, guardianship), person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient undergoing vitrectomy or preindentation in the ophthalmology department of Rennes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of the flare value | Changes between baseline (preoperatively) and day 7, month 1, month 2, month 3, month 6, and month 12 measures
  Evolution of the flare value preoperatively and then to D7, M1, M2, M3, M6, M12 of the operated eye

SECONDARY OUTCOMES:
Flare values of the fellow eye and the operated eye | Difference between flare values of the fellow eye and the operated eye at each evaluation time : baseline (preoperatively), day 7, month 1, month 2, month 3, month 6, and month 12
  Flare value of the fellow eye and the operated eye at each evaluation time

OTHER OUTCOMES:
Flare value of the operated eye | Changes between baseline (preoperatively) and day 7, month 1, month 2, month 3, month 6, and month 12 measures
  Flare value of the operated eye preoperatively and at each evaluation time
Criteria associated with high inflammation | Baseline (preoperatively)
  Identification of criteria associated with high inflammation : indication of surgery
Criteria associated with high inflammation | Baseline (preoperatively)
  Identification of criteria associated with high inflammation : ophthalmologic antecedents
Criteria associated with high inflammation | Baseline (preoperatively)
  Identification of criteria associated with high inflammation : high preoperative IOP
Criteria associated with high inflammation | Baseline (preoperatively)
  Identification of criteria associated with high inflammation : BCVA (better visual acuity corrected) preoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Dalal ASRI, Principal Investigator — Rennes University Hospital